CLINICAL TRIAL: NCT05979090
Title: Mastery Learning in Communication Skills to Improve Milestone Performance and Burnout
Brief Title: Mastery Learning in Communication Skills
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 20235952
Record Dates: First submitted 2023-07-19; First posted 2023-08-07 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Communication Research; Communication, Personal; Burnout, Professional
MeSH Terms: conditions — Communication; Burnout, Professional

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mastery Learning Group (Experimental)
  Interventions: Behavioral: Mastery learning in communication skills
- Standard of Care Group (No Intervention)

INTERVENTIONS:
Behavioral: Mastery learning in communication skills — Participants will undergo simulation-based mastery learning curriculum in difficult conversations.
  Arms: Mastery Learning Group

SUMMARY:
The goal of this study is to determine whether mastery learning in communication skills can improve skills in a simulated environment and have translational improvements in outcomes. The main questions it aims to answer are: 1. Does mastery learning improve skills in the simulation laboratory? 2. Does mastery learning improve clinical skills as seen by milestone performance? and 3 Does mastery learning improve burnout levels? The study is a multi-institutional randomized controlled trial of anesthesiology residents from five different residency programs. Participants will be randomized to mastery training in communication skills and standard of care, which is vicarious learning. Researchers will compare these two groups to see if mastery learning improves skills and translational outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Anesthesiology residents rotating at Ann and Robert H. Lurie Children's Hospital of Chicago

Exclusion Criteria:

* Participant refusal
* Study participants who have already undergone the mastery learning in difficult conversations course.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-01-18 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Communication skills | one year
  Post test checklist skills scores, a 16-item checklist was developed using the modified Delphi technique with possible scores of 0 (lowest) to 16 (highest). All items in the checklist are graded dichotomously and (1 if done correctly and 0 if not done or done incorrectly.

SECONDARY OUTCOMES:
Milestones Performance | two years
  The ACGME interpersonal and communication core competency is subdivided into three Anesthesiology Milestones: Patient and Family-centered communication, Interprofessional and Team Communication, and Communication within Health Care Systems. Each milestone is graded on a score of 1 (novice) to 5 (expert) by each residency program's Clinical Competency Committee (CCC).
Burnout levels | 1.5 years
  The Maslach Burnout Inventory Scale (MBI-9) will be used to estimate the levels of burnout prior to participation in the intervention, immediately after course completion, and at 2 and 6 months after training. The MBI is a measure of job burnout defined by three subscales: emotional exhaustion (EE) (9 items), depersonalization (DP) (5 items), and professional accomplishment (PA) (8 items), each with 7-point Likert-type, frequency response scale (0 = never, 1 = a few times a year or less, 2 = once a month or less, 3 = a few times a month, 4 = once a week, 5 = a few times a week, 6 = every day) [1, 2]. Scales are scored such that higher scores indicate more of each construct. Higher scores on the EE and DP subscales indicate a higher burnout symptom burden; lower scores on the PA subscale indicate a higher burnout symptom burden.

CONTACTS AND LOCATIONS:
Overall Officials: Heather Ballard, MD, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (1):
- Northwestern University Simulation Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
de-identified study data will be available upon request when study is completed and published